CLINICAL TRIAL: NCT06437366
Title: Effectiveness of a Nurse-Led Heart Math Training Program on Resilience , Sense of Coherence, and Emotional Adjustment in Patients With Substance Use Disorder
Brief Title: Nurse-Led Heart Math Training Program With Substance Use Disorder
Acronym: HeartMathsub
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 100.a
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nurse-led HeartMath training program on patients with substance use disorder (Experimental): The HeartMath training program, developed by the HeartMath Institute, focuses on teaching individuals self-regulation skills that promote heart-brain coherence. This state of coherence has been associated with improved cognitive function, emotional stability, and physical health. By integrating this training into the care of patients with SUDs, nurses can play a pivotal role in addressing the complex emotional and psychological needs of this population.
  Interventions: Behavioral: Nurse-Led Heart Math Training Program
- Non-experimental patients with substance use disorder (No Intervention)

INTERVENTIONS:
Behavioral: Nurse-Led Heart Math Training Program — he nurse-led HeartMath training program consists of several key components designed to enhance resilience, sense of coherence, and emotional adjustment:
  Heart-Focused Breathing Techniques: Patients are taught specific breathing techniques that help synchronize heart and brain activity, leading to a state of physiological coherence.
  Emotional Regulation Skills: The training includes exercises that help individuals recognize and shift from negative to positive emotional states, thereby improving emotional stability and reducing stress.
  Arms: nurse-led HeartMath training program on patients with substance use disorder

SUMMARY:
Substance use disorders (SUDs) pose significant challenges to individuals' psychological well-being, resilience, and emotional adjustment. These disorders often lead to detrimental effects on physical health, mental health, and overall quality of life, creating a critical need for effective interventions that can support recovery and enhance emotional resilience. One promising approach is the implementation of nurse-led HeartMath training programs. These programs utilize evidence-based techniques to improve emotional regulation, increase resilience, and foster a sense of coherence, which is the ability to perceive life as comprehensible, manageable, and meaningful.

DETAILED DESCRIPTION:
The HeartMath training program, developed by the HeartMath Institute, focuses on teaching individuals self-regulation skills that promote heart-brain coherence. This state of coherence has been associated with improved cognitive function, emotional stability, and physical health. By integrating this training into the care of patients with SUDs, nurses can play a pivotal role in addressing the complex emotional and psychological needs of this population.

Brief About the Training Program

The nurse-led HeartMath training program consists of several key components designed to enhance resilience, sense of coherence, and emotional adjustment:

Heart-Focused Breathing Techniques: Patients are taught specific breathing techniques that help synchronize heart and brain activity, leading to a state of physiological coherence.

Emotional Regulation Skills: The training includes exercises that help individuals recognize and shift from negative to positive emotional states, thereby improving emotional stability and reducing stress.

Biofeedback Technology: Participants use HeartMath biofeedback devices that provide real-time feedback on their heart rhythm patterns, enabling them to monitor and improve their coherence levels.

Resilience-Building Exercises: The program incorporates activities and practices aimed at enhancing personal resilience, such as positive visualization and the cultivation of gratitude and appreciation.

Individual and Group Sessions: The training is delivered through a combination of individual coaching and group workshops, providing both personalized support and a sense of community.

ELIGIBILITY:
Inclusion Criteria:

* substance abuse for at least one month

Exclusion Criteria:

* out side hospital

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Patients with substance use disorder who participate in a nurse-led HeartMath training program | three months
  Patients with substance use disorder who participate in a nurse-led HeartMath training program will show a statistically significant increase in resilience, as measured by the Connor-Davidson Resilience Scale (CD-RISC), compared to those who do not participate in the program.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Alexandria Governorate, Egypt

REFERENCES:
- [Derived] Elzohairy NW, Eweida RS, Othman AA, Hammad HA, Ramadan Atta MH. Effectiveness of a Nurse-Led HeartMath Training Program on Resilience, Emotional Adjustment, and Treatment Motivation Among Patients With Substance Use Disorder: A Randomized Control Trial. Worldviews Evid Based Nurs. 2025 Aug;22(4):e70061. doi: 10.1111/wvn.70061. PMID 40708166